CLINICAL TRIAL: NCT07285226
Title: Impact of 12-Week Creatine HCl Supplementation on Body Composition, Functional Muscle and Brain Performance, Blood Biomarkers, and Tissue Creatine Levels in Older Adults With Sarcopenia
Brief Title: Creatine HCl Supplementation in Sarcopenia: A Randomized Controlled Study
Acronym: SARCOPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4005-31-01
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1 (Experimental): 2 capsules of creatine HCl per day
  Interventions: Dietary Supplement: Experimental 1
- Experimental 2 (Placebo Comparator): 2 capsules of inulin HCl per day
  Interventions: Dietary Supplement: Experimental 2

INTERVENTIONS:
Dietary Supplement: Experimental 1 — Creatine HCl
  Arms: Experimental 1
Dietary Supplement: Experimental 2 — Innulin (placebo)
  Arms: Experimental 2

SUMMARY:
The CONCRET-SARCOPA trial is a 12-week, double-blind, randomized controlled study designed to evaluate the efficacy of creatine HCl supplementation in older adults with sarcopenia. The trial investigates whether daily creatine HCl improves body composition, enhances functional muscle and cognitive performance, and favorably alters key blood biomarkers associated with muscle health and metabolic status. Additionally, the study assesses changes in tissue creatine levels using non-invasive and biochemical methods to clarify mechanistic responses to supplementation. Findings from this trial will provide critical evidence on the therapeutic potential of creatine HCl as a targeted nutritional strategy for managing sarcopenia in the geriatric population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Low muscle strength by handgrip (SDOC criteria for sarcopenia): < 35.5 kg in men and < 20 kg in women
* Sign free and informed consent
* Demonstrate interest, conditions and availability to participate

Exclusion Criteria:

* Patients undergoing interventional treatment for sarcopenia
* Physical amputation
* Cognitive impairment (MSSE < 25)
* Unwillingness to return for follow-up analysis
* Participation in other clinical trials

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Hand-grip strength | Change from baseline hand-grip strength at 12 weeks
  Handgrip strength quantifies maximal voluntary force generated by the hand using a dynamometer, serving as a simple, reliable indicator of overall muscle function and sarcopenia severity.

SECONDARY OUTCOMES:
Senior fitness test score | Change from baseline senior fitness test score at 12 weeks
  The Senior Fitness Test score reflects aggregated performance across multiple functional tasks, providing a quantifiable index of an older adult's overall physical capability, mobility, and age-related fitness status.
Mini-Mental State Examination Score | Change from baseline Mini-Mental State Examination Score at 12 weeks
  The Mini-Mental State Examination score quantifies global cognitive function by assessing orientation, memory, attention, language, and visuospatial abilities, offering a validated measure for detecting cognitive decline in older adults.
Appendicular muscle mass | Change from baseline appendicular muscle mass at 12 weeks
  Appendicular muscle mass quantifies lean soft tissue in arms and legs serving as a key indicator of skeletal muscle quantity and sarcopenia-related muscle depletion.
Brain creatine | Change from baseline brain creatine concentrations at 12 weeks
  Magnetic resonance spectra for brain creatine concentrations
Irisin | Change from baseline serum levels of irisin at 12 weeks
  Serum levels of irisin

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Study Chair — Center for Mitochondrial Medicine
Locations (1):
- Center for Health Sciences, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in sarcopenia. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in perimenopause.

REFERENCES:
- [Background] Eghbali E, Arazi H, Suzuki K. Supplementing With Which Form of Creatine (Hydrochloride or Monohydrate) Alongside Resistance Training Can Have More Impacts on Anabolic/Catabolic Hormones, Strength and Body Composition? Physiol Res. 2024 Nov 15;73(5):739-753. doi: 10.33549/physiolres.935323. PMID 39545789
- [Background] Korovljev D, Ostojic J, Panic J, Ranisavljev M, Todorovic N, Nedeljkovic D, Kuzmanovic J, Vranes M, Stajer V, Ostojic SM. The Effects of 8-Week Creatine Hydrochloride and Creatine Ethyl Ester Supplementation on Cognition, Clinical Outcomes, and Brain Creatine Levels in Perimenopausal and Menopausal Women (CONCRET-MENOPA): A Randomized Controlled Trial. J Am Nutr Assoc. 2025 Aug 25:1-12. doi: 10.1080/27697061.2025.2551184. Online ahead of print. PMID 40854087
- [Background] Tuckfield C. First use of creatine hydrochloride in premanifest Huntington disease. Med J Aust. 2015 Apr 20;202(7):378-80. doi: 10.5694/mja14.01070. No abstract available. PMID 25877121